CLINICAL TRIAL: NCT05509946
Title: Preemptive Analgesia Combination of Celecoxib and Pregabalin in Total Hip Arthroplasty: Comparison of the Effects of Single Dose and Repeated Doses (Double-Blind Randomized Clinical Trial)
Brief Title: Preemptive Analgesia Combination of Celecoxib and Pregabalin in THA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kemas Muhammad Azka Novriandi, Medical doctor, Orthopaedic Surgeon, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID2564
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Arthroplasty Complications; Analgetic; Celecoxib; Pregabalin
Keywords: total hip arthroplasty; celecoxib; pregabalin; preemptive analgetic
MeSH Terms: interventions — Celecoxib; Pregabalin

STUDY DESIGN:
Intervention Model Description: There are 3 separate groups defined by randomization:
  1. single dose of combined celecoxib 400 mg and pregabalin 150 mg an hour before surgery
  2. repeated dose of combined celexocib 200 mg twice a day and pregabalin 75 mg twice a day, administered 3 days before surgery
  3. placebo administered an hour before surgery
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization performed by simple random sampling, the result is latern given to investigator in an envelope containing codes made by third party outside the research. Investigator and the patient do not know the allocation code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose of celecoxib 400 mg and pregabalin 150 mg (Experimental): Single dose of celecoxib 400 mg and pregabalin 150 mg administered an hour before surgery
  Interventions: Drug: Single dose of celecoxib 400 mg and pregabalin 150 mg
- Repeated dose of celecoxib 200 mg and pregabalin 75 mg (Active Comparator): Repeated dose of celecoxib 200 mg twice a day and pregabalin 75 mg twice a day administered starting from 3 days before surgery
  Interventions: Drug: Repeated dose of celecoxib 200 mg and pregabalin 75 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Single dose of celecoxib 400 mg and pregabalin 150 mg — Single dose of celecoxib 400 mg and pregabalin 150 mg
  Arms: Single dose of celecoxib 400 mg and pregabalin 150 mg
Drug: Repeated dose of celecoxib 200 mg and pregabalin 75 mg — Repeated dose of celecoxib 200 mg and pregabalin 75 mg started 3 days before surgery
  Arms: Repeated dose of celecoxib 200 mg and pregabalin 75 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded randomized controlled trial aims to evaluate the effect of preemptive analgetic combination of celecoxib and pregabalin to acute pain after total hip arthroplasty. This study will be conducted in Cipto Mangunkusumo Hospital, Jakarta, Indonesia, from October 2022 to April 2023. The subject of this study is adult patient who will be performed total hip arthroplasty.

DETAILED DESCRIPTION:
1. Research design This is a double-blind, randomized clinical trial which aimed to evaluate the effect of preemptive analgesia combined with Celecoxib and Pregabalin on acute post-THA pain.
2. Study location This study will be conducted at the Cipto Mangunkusumo Hospital, Jakarta, Indonesia.
3. Study time This study will be conducted in October 2022 - April 2023
4. Population and sample The target population of this study is adult patients undergoing THA surgery. The randomization technique used in this study is a simple randomization technique. Researchers randomly determine the allocation of samples without looking at subjects' status in the population.
5. Inclusion criteria

   * Patients >18 years old
   * Patients who come to the RSCM Orthopedic Polyclinic
   * Patients undergoing THA surgery
   * Patients with Primary and Secondary Pelvic Osteoarthritis
   * The patient is taking anti-pain and anti-inflammatory drugs regularly
6. Exclusion criteria

   * Patients with mental disorders
   * Patients with a history of renal impairment
   * Pelvic arthritis patients due to rheumatoid arthritis or infection
   * Patients with diabetes and obesity
   * Allergy to non-steroidal inflammatory drugs
   * Asthma history
   * Coagulation disorders
   * Patients in the study procedure experienced an incident of severe pain that required another analgesic regimen
   * History of hypersensitivity to NSAIDs or sulfonamides

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old
2. Patients who come to the RSCM Orthopedic Polyclinic
3. Patients undergoing THA operasi surgery
4. Patients with Primary and Secondary Pelvic Osteoarthritis
5. The patient is taking anti-pain and anti-inflammatory drugs regularly

Exclusion Criteria:

1. Patients with mental disorders
2. Patients with a history of renal impairment
3. Pelvic arthritis patients due to rheumatoid arthritis or infection
4. Patients with diabetes and obesity
5. Allergy to non-steroidal inflammatory drugs
6. Asthma history
7. Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | After surgery for three days
  Acute pain measured in the morning before activity after surgery. Measured by numeric pain rating scale 0 - 10 which lower score means less pain while higher score means more pain
Total consumption of morphine | Three days
  Morphine is an opioid analgesic, in this study it was used as an analgesic as well as an objective parameter to assess the effectiveness of celecoxib and pregabalin. Given with a patient control analgesia (PCA) device. Dosage of morphine used

CONTACTS AND LOCATIONS:
Overall Officials: Andri MT Lubis, Study Director — Department of Orthopaedic and Traumatology, Faculty of Medicine, Universitas Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathappan SS, Strauss EJ, Ginat D, Upasani V, Di Cesare PE. Surgical challenges in complex primary total hip arthroplasty. Am J Orthop (Belle Mead NJ). 2007 Oct;36(10):534-41. PMID 18033565
- [Background] Boisgard S, Descamps S, Bouillet B. Complex primary total hip arthroplasty. Orthop Traumatol Surg Res. 2013 Feb;99(1 Suppl):S34-42. doi: 10.1016/j.otsr.2012.11.008. Epub 2013 Feb 1. PMID 23375960
- [Background] Ferrata P, Carta S, Fortina M, Scipio D, Riva A, Di Giacinto S. Painful hip arthroplasty: definition. Clin Cases Miner Bone Metab. 2011 May;8(2):19-22. PMID 22461810
- [Background] Arden NK, Kiran A, Judge A, Biant LC, Javaid MK, Murray DW, Carr AJ, Cooper C, Field RE. What is a good patient reported outcome after total hip replacement? Osteoarthritis Cartilage. 2011 Feb;19(2):155-62. doi: 10.1016/j.joca.2010.10.004. Epub 2010 Oct 15. PMID 20951814
- [Background] Hayes JH, Cleary R, Gillespie WJ, Pinder IM, Sher JL. Are clinical and patient assessed outcomes affected by reducing length of hospital stay for total hip arthroplasty? J Arthroplasty. 2000 Jun;15(4):448-52. doi: 10.1054/arth.2000.4346. PMID 10884204
- [Background] Holtzman J, Saleh K, Kane R. Effect of baseline functional status and pain on outcomes of total hip arthroplasty. J Bone Joint Surg Am. 2002 Nov;84(11):1942-8. doi: 10.2106/00004623-200211000-00006. PMID 12429753
- [Background] Pinto PR, McIntyre T, Araujo-Soares V, Costa P, Ferrero R, Almeida A. A comparison of predictors and intensity of acute postsurgical pain in patients undergoing total hip and knee arthroplasty. J Pain Res. 2017 May 9;10:1087-1098. doi: 10.2147/JPR.S126467. eCollection 2017. PMID 28533697
- [Background] Singh JA, Noorbaloochi S, Knutson KL. Cytokine and neuropeptide levels are associated with pain relief in patients with chronically painful total knee arthroplasty: a pilot study. BMC Musculoskelet Disord. 2017 Jan 14;18(1):17. doi: 10.1186/s12891-016-1375-2. PMID 28088207